CLINICAL TRIAL: NCT04110353
Title: Prophylactic Closed Incision Negative Pressure Wound Therapy on Abdominal Wounds - Clinical and Economic Perspectives: A Multi-centre Randomised Trial
Brief Title: Prophylactic Closed Incision Negative Pressure Wound Therapy on Abdominal Wounds - Clinical and Economic Perspectives
Acronym: ProNounCE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 19IC5400
Record Dates: First submitted 2019-09-20; First posted 2019-10-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Wound Infection; Surgical Site Infection; Surgical Wound; Surgical Incision
Keywords: Surgical Site infections; Negative Pressure Wound Therapy; Contaminated abdominal wounds; Closed incision abdominal wound; Prophylactic therapy
MeSH Terms: conditions — Wound Infection; Surgical Wound Infection; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Stepped wedge design with randomisation at the level of the Hospitals not individual patients
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative dressings (Active Comparator): Use of simple dressings on wound post operatively - to be placed at end of operation
  Interventions: Other: Wound dressings: Conservative dressings
- Prevena dressing (Active Comparator): Use of Prevena(KCI) dressing on wound post operatively - to be placed at end of operation
  Interventions: Other: Wound dressings: Prevena dressings
- ciVAC dressing (Active Comparator): Use of closed incision VAC (vacuum assisted closure) dressing on wound post operatively - to be placed at end of operation
  Interventions: Other: Wound dressings: ciVAC dressings

INTERVENTIONS:
Other: Wound dressings: Conservative dressings — Conservative dressings to be placed on closed wounds post operatively, after open operations on the bowel. To be changed at day 7 or sooner if clinically indicated.
  Arms: Conservative dressings
Other: Wound dressings: Prevena dressings — Prevena dressing to be placed on closed wounds post operatively, after open operations on the bowel. To be changed at day 7 or sooner if clinically indicated.
  Arms: Prevena dressing
Other: Wound dressings: ciVAC dressings — Closed incision VAC dressings to be placed on closed wounds post operatively, after open operations on the bowel. To be changed at day 7 or sooner if clinically indicated.
  Arms: ciVAC dressing

SUMMARY:
This study evaluates whether specialist negative pressure dressings reduce the risk of wound infections after operations when compared to conservative dressings, and if one negative pressure dressings works better than another. The study will look at patients who have had an open operation on their bowel and the wound closed at the end of the operation.

DETAILED DESCRIPTION:
Surgical site infections (SSI) can affect up 41% of patients post-operatively. They are associated with significant healthcare and patient costs, and increased patient morbidity and mortality.

Specialist post operative dressings with negative pressure wound therapy are available, and the WHO do recommended for use in high risk wounds, taking resources into account. However no further recommendations are available.

This study will explore the rate of post-operative wound infections in adult patients undergoing open abdominal surgery on the bowel, and compare the rate of wound infections in these patients in relation to three different dressing types used after their operation. The study aims to determine if any of the dressings used within the study are associated with lower post-operative wound infection rates, and compare the overall costs of using each dressing type, including both direct healthcare costs and societal costs. Finally, it will evaluate participant's quality of life outcomes after open abdominal surgery, specifically relating to their wound.

ELIGIBILITY:
Inclusion Criteria:

* Emergency, trauma or elective contaminated abdominal operations within general surgery and/or colorectal surgery
* Abdominal wounds closed at time of operation and expected to heal by primary intention
* Patients who have the capacity to consent
* To include complex abdominal wounds with existing infection where wounds have been closed and expected to heal by primary intention
* To including graft or flap sites as part of general surgical procedure
* Patients who are able to complete questionnaires post operatively, either alone or with assistance

Exclusion Criteria:

* Wounds where an appropriate seal cannot be obtained
* Wounds left open and expected to heal by secondary intention
* Patients known to have allergy or sensitivity to dressings being used
* Patients who lack the capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | Up to day 90
  The occurrence of surgical site infections at the post-operative wound and timeframe of occurrence

SECONDARY OUTCOMES:
Wound assessments - clinical assessment of presence of wound complication and healing | At day 7 (on removal of dressing), up to day 30 (on discharge), day 40 (at outpatient follow up)
  Independent blind assessment of wounds at day 7 post operatively, on discharge and at outpatient follow up, via wound photographs taken, and correlation with assessment by clinical team
Length of stay | Up to 90 days
  Length of stay post-operatively
Number of additional interventions received by participants due to development of a Surgical Site Infection | Within 30 days
  Need for intervention or treatment for surgical site infection (antibiotics, opening up of wound at bedside, operative or radiological intervention)
Microscopy, culture and sensitivity results from swabs of any Surgical Site Infections | Within 30 days
  Culture results if SSI post-operative (including sensitivities)
Post operative complications - other | Within 30 days
  Occurrence of other post-operative complications
Number of adverse reactions to treatments for Surgical Site Infections | Within 30 days
  Adverse reactions to antibiotics given or to dressings use
Wound dressings - use of | Up to day 30-40
  Time to discontinuation of dressings, type and number of dressings used
Ninety day mortality rate | Up to day 90
  Mortality within 90 days
Ninety day readmission rate | Up to day 90
  Rate of readmission within 90 days
Cause of death | Up to day 90
  Cause of death for any mortalities within 90 days
Quality of life measures: EuroQol 5 Dimensions 5 Levels (EQ5D5L) questionnaire | At day 7 (on removal of dressing), up to day 30 (on discharge), day 40 (at outpatient follow up)
  Generic quality of life outcome measures using EQ5D5L questionnaire assessed at day 7 post operatively, on discharge and at outpatient follow up; individualised questions, no formal scale
Quality of life measures: Wound Quality of Life questionnaires | At day 7 (on removal of dressing), up to day 30 (on discharge), day 40 (at outpatient follow up)
  Wound specific quality of life outcome measures using Wound Quality of Life questionnaire assessed at day 7 post operatively, on discharge and at outpatient follow up; scales - not at all/a little/moderately/quite a lot/very much
Quality of life and economic measures: Economic assessment questionnaire | At day 40
  Assessment of economic impact of wound using single Economic questionnaire to be assessed at day 40; individualised questions that will be assessed, no formal scale
Long term follow up - Hernia occurrence | At 1, 3 and 5 years
  Development of incisional hernia

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Peters, Principal Investigator — Imperial College London; Carolynne Vaizey, Study Chair — St Mark's Hospital and Academic Institute

IPD SHARING:
Plan to Share IPD: No